CLINICAL TRIAL: NCT04808518
Title: An Observational Primary Data Collection Study to Compare the Lung Function in the Adult Severe Asthma Patients Who Start Biologics Treatment and Who do Not Start, After Two-year Follow-up
Brief Title: A Study to Compare Severe Asthma Patients Who Start Biologics and Who do Not Start (PROSPECT)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00062
Record Dates: First submitted 2021-03-05; First posted 2021-03-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Bx reg group
- non-Bx reg group

SUMMARY:
Objectives in this study is to compare the change of lung function after 24 months from baseline between the two groups; one is the patient group who decided to start biologics treatment, and another is the patient group who decided to start non-biologics treatment. The target patients are the adult uncontrolled severe asthma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed asthma diagnosis
2. Using high-dose ICSa and 2nd controllerb more than 3 months before registration
3. Uncontrolled asthma which constitutes one or more of 1) Poor symptom control: ACQ-5≧1.5 or ATC<20 2) Frequent exacerbations: at least 2 asthma exacerbations in the 12 months prior to the registration 3) Airflow obstruction: FEV1 before taking bronchodilator <80% predicted (FEV1/FVC less than the lower limit of normal) C
4. Investigators judges the necessity of biologic treatment for his/her asthma treatment and the patients are explained the situation by the investigators.
5. Patients deemed capable of visiting their study site next 24 months regularly
6. Patients from whom written consent to participate in this study has been obtained
7. Patients≧20 years old at obtaining consent

Exclusion Criteria:

1. Participated in other interventional studies such as clinical trials, etc within the last 8 weeks.
2. Are using biologics at registration
3. Diagnosed as COPD
4. Plan the BT therapy near future
5. Receipt of any marketed or investigational biologics within 5 months before the registration
6. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target patients in this study are the adult severe asthma patients whose asthma control status is uncontrolled based on the definition of ERS/ATS guideline. Also, the investigators judge the necessity of biologic treatment and explain the situation to these patient population.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Post-bronchodilator Forced Expiratory Volume in 1 Second (Post-BD FEV1) | 24 months from baseline
  Change from baseline in post-bronchodilator Forced Expiratory Volume in 1 Second (Post-BD FEV1) at 24 months

SECONDARY OUTCOMES:
Changes in Post-BD FEV1 | Until 24 months from baseline
  To describe the value of lung function decline in Bx reg and non-Bx reg by changes in Post-BD FEV1 from 6 months to 24 months, and from 12 months to 24 months
Post-BD FEV1 by patient's background | Until 24 months from baseline
  Change from baseline in post-bronchodilator FEV1 at 24 months by patient's background,
  To compare the differences of change from baseline in post-BD FEV1 at 24 months between Bx reg and non-Bx reg, by the following patients' sub-groups
  1. Number of exacerbations during the study period (0, 1-2, 3-4, >= 5)
  2. asthma control level (mean ACQ-5 score between 6 months and 24 months; <0.75, 0.75 - 1.5, >1.5)
To compare the asthma control status between Bx reg and non-Bx reg | 24 months from baseline
  To compare the asthma control status during the study period (24 months) between Bx reg and non-Bx reg -ACQ-5,Time to first asthma exacerbation and so on
Daily Oral Corticosteroid use | Until 24 months from baseline
  Change from baseline in daily Oral Corticosteroid dose, Time to withdraw regular Oral Corticosteroid use
Baseline patient background and clinical presentations between Bx reg and non-Bx reg | Until 24 months from baseline
  To describe the baseline patient background and clinical presentations between Bx reg and non-Bx reg
MiniAQLQ score | Until 24 months from baseline
  To compare the differences of change from baseline in MiniAQLQ score between both groups at 24 months
ACQ-5 score | 24 months from baseline
  To compare the differences of change from baseline in ACQ-5 score at 12 months and 24 months between both groups.
  To compare the asthma control status during the study period (24 months) between Bx reg and non-Bx reg by ACQ-5 score.
Time to first asthma exacerbation | 24 months from baseline
  To compare the asthma control status during the study period (24 months) between Bx reg and non-Bx reg by Time to first asthma exacerbation
Annual rate of asthma exacerbations | 24 months from baseline
  To compare the asthma control status during the study period (24 months) between Bx reg and non-Bx reg by Annual rate of asthma exacerbations
Asthma-specific resource utilisation (Hospital visits, ER/urgent care visits, hospitalisations) | 24 months from baseline
  To compare the asthma control status during the study period (24 months) between Bx reg and non-Bx reg by Asthma-specific resource utilisation (Hospital visits, ER/urgent care visits, hospitalisations)

OTHER OUTCOMES:
To describe baseline patients' background and clinical presentations by each biologic | Until 24 months from baseline
  To describe baseline patients' background and clinical presentations by each biologic - Age, sex, , BMI, smoking history, history of pediatric asthma, duration of asthma, complications, comorbidities, blood eosinophils, FeNO, IgE, Atopic factor, etc.
Blood eosinophil counts, FeNO, Atopic factor, IgE in non-Bx reg | Until 24 months from baseline
  To describe the proportion of these patient population in non-Bx reg; Blood eosinophil counts, FeNO, Atopic factor, IgE in non-Bx reg
Time to decrease 0.5 (at least) of ACQ-5 score and duration of asthma | Until 24 months from baseline
  To evaluate the association between the time to decrease 0.5 of ACQ-5 and duration of asthma (< 10 years, 10<= and < 20 years, 20<= and < 30 years, >= 30 years)
Treatment reality of each biologic | Until 24 months from baseline
  To describe the following information in Bx reg during the observational period
  * Reason why a biologic is switched to another biologic
  * Time to switch the biologic
  * Specific biologic at the first time, at the 2nd time, etc.
  * Chronological change of proportion of prescribed each biologic during the observational period
To describe the change of asthma control status after switching one biologic to other biologics by ACQ-5 score status | Until 24 months from baseline
  To describe the change of asthma control status after switching one biologic to other biologics by the following ACQ-5 score status
  * ACQ-5 responder rate (respond; decrease of more than 0.5 score)
  * Proportion of the following category by ACQ-5 score change pre/post switching (improve: -0.5 =<, no-change: -0.5< ACQ-5 <0.5, worse: >=0.5)
To explore the factors related to non-responder in Bx reg group | Until 24 months from baseline
  To explore the factors related to non-responder at 24 months in Bx reg group (Definition of non-responder; ACQ-5 score decrease from the baseline is no more than 0.5[<0.5] )
Reason why biologics are not started within 12 weeks in non-Bx reg group | within 12 weeks from study start
  To describe the reason why biologics are not started within 12 weeks in non-Bx reg group.

CONTACTS AND LOCATIONS:
Locations (28):
- Japan (28):
  - Research Site, Aki-gun Fucyu
  - Research Site, Asahikawa
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Ikoma
  - Research Site, Kobe
  - Research Site, Kumagaya
  - Research Site, Maebashi
  - Research Site, Meguro City
  - Research Site, Nagoya
  - Research Site, Nangōku
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōtsu
  - Research Site, Sagamihara
  - Research Site, Sayama
  - Research Site, Shinagawa City
  - Research Site, Shinjuku
  - Research Site, Shizuoka
  - Research Site, tabashi City
  - Research Site, Toyoake
  - Research Site, Tsukubo-gun Hayashima
  - Research Site, Yamagata
  - Research Site, Yokohama
  - Research Site, Yonago

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00062&attachmentIdentifier=9f4f82fd-c600-4359-8c06-474982d32d26&fileName=PROSPECT_CSR_Final_03Jul2024_Synopsis.pdf&versionIdentifier=